CLINICAL TRIAL: NCT03143322
Title: Extracranial Stereotactic Body Radiation Therapy (SBRT) Added to Standard Treatment Versus Standard Treatment Alone in Solid Tumors Patients With Between 1 and 5 Bone-only Metastases
Brief Title: Standard Treatment +/- SBRT in Solid Tumors Patients With Between 1 and 5 Bone-only Metastases
Acronym: STEREO-OS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UC-0107/1603
Record Dates: First submitted 2017-04-28; First posted 2017-05-08 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Breast Cancer; Metastatic Lung Cancer; Metastatic Prostate Cancer; Bone Metastases
Keywords: Bone-only metastases; solid tumors; SBRT
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms; Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Systemic treatment + SBRT (Experimental): Systemic treatment and SBRT to the bone metastases. Two SBRT schemes are allowed: 9 Gy x 3 fractions or 7 Gy x 5 fractions for axial and appendicular bones metastases. The choice is at the discretion of the investigator.
  Interventions: Radiation: SBRT
- Systemic treatment (No Intervention): Palliative radiotherapy on bone metastases is allowed if necessary (pain, fracture, spinal cord compression…)

INTERVENTIONS:
Radiation: SBRT — SBRT will be added to systemic (standard) treatment of bone metastases.
  Arms: Systemic treatment + SBRT

SUMMARY:
Bone metastases occur frequently during the evolution of solid tumors, either isolated or associated with visceral metastases. The incidence varies between 20 and 85% depending on the primary cancer. Breast, prostate, and lung cancers are responsible for 70% of bone metastases. Cancer with bone metastases compared to other metastatic sites is considered as associated with a better prognosis, particularly for breast and prostate cancer. Bone metastases may be present at diagnosis (synchronous metastasis) or appear at a later time (metachronous metastasis).

The concept of "oligometastases" was proposed in patients with about 3 up to 5 metastases (without restriction on the primary site) and associated with an intermediate prognosis. It was hypothesized that local treatment with curative intent, aiming at the few metastatic sites, would yield long-term survival probabilities, along with systemic therapies.

Long-term survivors have been reported after curative-intent treatment of metastasis in sarcoma and colorectal cancers with liver or lung metastasis. We chose to focus on bone metastasis because of their high incidence, their impact on the patient's quality of life and autonomy, and their accessibility to potentially curative radiotherapy.

The systemic treatment of metastatic cancer includes hormonal therapy (breast and prostate cancer), biologically-targeted drugs and chemotherapy (all cancers).

Stereotactic radiotherapy is a highly accurate technique was initially developed for performing the radiosurgery of brain tumors in patients for whom it was deemed be too difficult to proceed to classical excision surgery. In this process, a high total dose of radiation is delivered in a single fraction to a well-defined intra-cranial target. The concept of radiotherapy in stereotactic conditions was extended to one or several fractions delivered to small volumes primary tumors/ metastases in extra-cranial sites (Stereotactic Body RadioTherapy [SBRT]). At present, high control rates have been achieved for lung metastases. Similarly, very high local control rates have been reported in bone metastases after stereotactic radiotherapy.

In this protocol, our purpose is to demonstrate, via a randomized phase III trial, that high doses of radiotherapy, delivered in stereotactic conditions to the bone metastases (between 1 and 5 metastases) in solid tumor patients is able to improve the survival without progression.

ELIGIBILITY:
Inclusion Criteria:

1. Patients older than 18 years and younger than 75 years
2. Good general condition: WHO performance status ≤ 2
3. Patients with histological proof of breast, non-small cell lung, or prostate cancer Note: Histological proof can be done on the primitive tumour and/or adenopathy and/or metastatic site.
4. Absence of co-morbidity contra-indicating radio-chemotherapy or surgery
5. Primary tumor accessible to curative-intent treatment (surgery, chemoradiation…) for patients with synchronous metastases
6. Patients with between 1 and 5 synchronous or metachronous bone metastases as defined by NaF-PET or conventional SPECT-CT scan and spinal MRI (if necessary) within 6 weeks before randomization)
7. Bones metastases treatable by SBRT
8. Primary cancer considered to be controlled or accessible to curative-intent treatment (surgery, chemoradiation…) in case of locoregional recurrence for metachronous bone oligo-metastatic disease
9. Women of childbearing potential and male patients must agree to use adequate contraception for the duration of study participation and up to 3 months following completion of therapy
10. Patients who have received the information sheet, dated and signed the informed consent form
11. Affiliated to the social security system

Exclusion Criteria:

1. Visceral metastases as defined by FDG-PET (F-Choline-PET or PSMA PET-CT for prostate cancer) and cerebral CT or MRI performed.
2. Previous systemic therapy for metastasis for patients with metachronous metastasis. Prostate and breast cancer patients remain eligible if hormonal treatment was initiated 6 months before enrollment
3. All bone metastasis requiring surgical treatment (spinal cord compression, fracture…)
4. More than 5 bone metastases as defined by NaF-PET or conventional SPECT-CT scan and spinal MRI (if spinal bone metastases on NaF-PET)
5. Previous cancer within the 5 years before inclusion (except basal cell carcinoma of the skin, in situ carcinoma of the uterine cervix)
6. Previous radiotherapy on bone metastasis (e.g: antalgic radiotherapy)
7. Patient enrolled in another therapeutic trial
8. Pregnant women or breast feeding mothers,
9. Hypersensitivity to the active substance (FDG and NaF or F-Choline or PSMA for prostate cancer) or to any of the excipients
10. Contraindication to MRI (in case of spinal metastases)
11. Patients deprived of liberty or placed under the authority of a tutor. Patients with any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial. Patients unable to understand the purpose of the study (language, etc.).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2018-07-24 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | 1 year
  To evaluate the impact of SBRT on Progression-Free Survival (PFS) at 1 year according to RECIST 1.1 and PERCIST 1.0 Criteria

SECONDARY OUTCOMES:
PFS at 2 and 3 years | 2 years and 3 years after treatment
  Progression-Free Survival (PFS) at 2 and 3 years will be evaluated according to RECIST 1.1 and PERCIST
Bone progression free survival at 1, 2 and 3 years | 1, 2 and 3 years after treatment
  Distant bone progression at 2 and 3 years will be evaluated according to RECIST Criteria 1.1 and at 1 year according to RECIST Criteria 1.1 and PERCIST
Local control at 1, 2 and 3 years | 1, 2 and 3 years after treatment
  Local control will be evaluated at 1, 2 and 3 years according to RECIST Criteria 1.1 and PERCIST
Cancer-specific survival | 1, 2 and 3 years after treatment
  The length of time from the start of treatment for the disease until the death identified as being due to the specified cancer.
Overall survival | 1, 2 and 3 years after treatment
  The length of time from the start of treatment for the disease until patients are still alive.
SBRT toxicities | 1, 2 and 3 years after treatment
  according CTCAE 4.0 scale
Patient's Quality of life | at baseline, 6 weeks after randomization, and 3 months, 6 months and 1, 2 and 3 years after treatment
  self-administered questionnaire
Pain score | at baseline, once a week during 2 weeks and 6 weeks after randomization, and at 3 months, 6 months and 1, 2 and 3 years after treatment
  according to Numeric Scale related to pain medication
Cost utility | 6 weeks after randomization
  QALYs (Quality-Adjusted Life Years) and ICERs (Incremental Cost-Effectiveness Ratios) calculation based on EQ-5D-3L questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastien Thureau, MD, Principal Investigator — Centre Henri Becquerel; Jean-Christophe Faivre, MD, Principal Investigator — Institut de Cancérologie de Lorraine - Alexis Vautrin
Locations (28):
- France (28):
  - ICO - Site Paul Papin, Angers
  - Centre Marie Curie, Arras
  - Hôpital Privé Les Bonnettes, Arras
  - Institut Sainte Catherine, Avignon
  - Centre Pierre Curie, Beuvry
  - Clinique Ambroise Pare, Beuvry
  - Clinique Tivoli Ducos, Bordeaux
  - Institut Bergonié, Bordeaux
  - Hôpital Métropole Savoie, Chambéry
  - Pôle Leonard de Vinci, Chambray-lès-Tours
  - Centre Amethyst CROM, Creil
  - Hôpital Henri Mondor, Créteil
  - Centre Léonard de Vinci, Dechy
  - Institut de Cancérologie de Bourgogne, Dijon
  - Chu Grenoble, Grenoble
  - Centre Oscar Lambret, Lille
  - Hôpital Privé Le Bois, Lille
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Centre de Cancérologie du Grand Montpellier, Montpellier
  - Institut de Cancérologie de Lorraine, Nancy
  - Institut de Cancérologie de l'Ouest, Nantes
  - Centre Catalan D'Oncologie, Perpignan
  - Institut Jean Godinot, Reims
  - Centre Henri Becquerel, Rouen
  - Centre d'oncologie et radiothérapie Saint-Jean, Saint-Doulchard
  - GCS RISSA - Institut de cancérologie Paris Nord, Sarcelles
  - Clinique des dentellières, Valenciennes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thureau S, Marchesi V, Vieillard MH, Perrier L, Lisbona A, Leheurteur M, Tredaniel J, Culine S, Dubray B, Bonnet N, Asselain B, Salleron J, Faivre JC. Efficacy of extracranial stereotactic body radiation therapy (SBRT) added to standard treatment in patients with solid tumors (breast, prostate and non-small cell lung cancer) with up to 3 bone-only metastases: study protocol for a randomised phase III trial (STEREO-OS). BMC Cancer. 2021 Feb 4;21(1):117. doi: 10.1186/s12885-021-07828-2. PMID 33541288